CLINICAL TRIAL: NCT07257471
Title: Application Research of Methylation Markers in Early-stage Lung Cancer Patients Treated With Co-ablation System Therapy
Status: Recruiting | Type: Observational
Sponsor: Beijing Haidian Hospital (Other)
Responsible Party: Principal Investigator, Yuqing Huang, Director, Beijing Haidian Hospital
Other Study IDs: M202552
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer (NSCLC)
Keywords: Liquid biopsy; ctDNA; Methylation biomarker; Prognostic monitoring; MRD; Co-ablation system therapy; Therapeutic efficacy evaluation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Co-ablation system therapy group: Lung cancer patients are treated with Co-ablation system therapy

SUMMARY:
Lung cancer has the highest global incidence and mortality among malignancies. While surgery is the primary curative treatment for early-stage patients, approximately 25-35% are ineligible due to comorbidities. For these patients, Co-ablation system therapy is a key minimally invasive option. However, even after imaging indicates complete tumor removal ("tumor-free status"), minimal residual disease (MRD) may persist, leading to recurrence.

Current mainstream MRD detection relies on identifying mutations in circulating tumor DNA (ctDNA). This approach faces challenges like high mutational heterogeneity and the frequent need for tumor tissue sequencing (Tumor-informed). In contrast, DNA methylation markers offer advantages: they do not require prior knowledge of tumor mutations, appear early in tumorigenesis, are tissue-specific, and allow sensitive detection via multiple consistent CpG sites. Recent studies confirm that ctDNA methylation-based MRD detection can predict recurrence in lung and colorectal cancers earlier than imaging and effectively stratify patient risk.

This study aims to investigate the role of SHOX2 and PTGER4 genes in plasma, for monitoring MRD and evaluating therapeutic efficacy in lung cancer patients after Co-ablation system therapy. The study will enroll non-small cell lung cancer (NSCLC) patients undergoing Co-ablation system therapy. Peripheral blood will be collected at multiple timepoints (pre-treatment up to 24 months post-treatment) for ctDNA methylation analysis. The correlation between methylation levels and radiological findings will be assessed. The predictive power for recurrence will be evaluated using ROC curves. Patients will be stratified into high-risk and low-risk groups based on methylation status. Kaplan-Meier survival analysis and Cox regression models will compare recurrence-free survival between groups and evaluate the independent predictive value of SHOX2/PTGER4 methylation for recurrence risk, providing a scientific basis for personalized treatment decisions and recurrence prediction.

DETAILED DESCRIPTION:
Lung cancer is one of the major malignant tumors threatening human life and health, with its incidence and mortality rates consistently ranking first among all malignant tumors globally. China has a high incidence of lung cancer. According to the latest data released by the National Cancer Center, in 2022, there were 1,060,600 new cases of lung cancer in China, accounting for 22.0% of all new malignant tumor cases, and 733,300 deaths, accounting for 28.5% of all malignant tumor deaths.

Among patients with non-small cell lung cancer (NSCLC), the risk of recurrence varies significantly across different stages: the 5-year recurrence rates are 19% for stage IA, 30% for stage IB, and 48.6% for stage II, while the 3-year recurrence rate for stage III patients is as high as 52%. Early surgical resection is the primary treatment method to improve the survival rate of lung cancer patients. As a local treatment modality, Co-ablation system therapy are particularly suitable for patients who cannot tolerate surgery or are ineligible for surgical treatment. However, postoperative recurrence and metastasis remain the core challenges in lung cancer treatment. Even when imaging examinations show that the tumor has achieved a so-called "no evidence of disease" status (R0 resection)-meaning the tumor has disappeared at the macroscopic and imaging levels-minimal residual disease (MRD) that may trigger cancer recurrence could still be hidden beneath this appearance.

Currently, mainstream MRD detection methods on the market rely on the detection of mutations in circulating tumor DNA (ctDNA). However, such mutation-based MRD detection has obvious limitations. For instance, the heterogeneity of tumor mutations among different patients is extremely high, making it difficult for small-sized detection panels to cover a broader patient population. The Tumor-inform detection approach achieves MRD detection by customizing a specific panel for each patient, but this method requires obtaining the patient's tumor tissue sample for sequencing, which to some extent limits its clinical application.

In contrast, when DNA methylation markers are used for MRD detection, there is no need to pre-obtain characteristic mutation information of the primary tumor, and the detection sensitivity is not affected by the number of high-frequency mutations in the patient's tumor. Moreover, DNA methylation modifications usually occur in the early stages of tumorigenesis and exhibit tissue specificity and cancer type specificity. At the same time, DNA methylation often maintains good consistency across multiple gene regions; therefore, MRD analysis can be achieved by detecting the methylation status of multiple CpG sites.

This study selected patients diagnosed with non-small cell lung cancer through histopathology or clinical diagnosis, all of whom underwent Co-ablation system therapy. Peripheral blood samples were collected from all enrolled patients at 3 days, 1 month, 3 months, 6 months, 12 months, 18 months, and 24 months after treatment for SHOX2/PTGER4 gene methylation detection. The study aims to explore whether this gene methylation detection can serve as an effective indicator for dynamic MRD monitoring in lung cancer patients after Co-ablation system therapy and to analyze its clinical efficacy in lung cancer patients. It is expected to provide a scientific basis for predicting the risk of lung cancer recurrence and guiding individualized treatment decisions, thereby avoiding overtreatment or delayed treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with non-small cell lung cancer by histopathology/clinical diagnosis; assessed by MDT as not suitable or refusing open or thoracoscopic resection surgery.
* Age 18-85 years old, gender unrestricted.
* The maximum diameter of the tumor is ≤ 5 cm (peripheral type) or ≤ 3 cm (central type), and the distance from major blood vessels/trachea is ≥ 1 cm.
* Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1, with an expected survival period of ≥ 6 months.
* The subjects should have clear case information, including age, gender, and clinical diagnosis, etc.

Exclusion Criteria:

* Those with a history of other malignant tumors or autoimmune diseases。
* Pregnant or lactating women; or patients with lung cancer who were negative for methylation before treatment.
* Patients with clinical or pathological diagnosis of lung metastatic cancer.
* Ppatients with multiple nodules and the current treatment cannot completely address all positive nodules.
* Patients whose clinical information or follow-up during the study may not be completed; and other factors that the researcher deems unsuitable for participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer (NSCLC) diagnosed by histopathology/clinical diagnosis and scheduled for Co-ablation system therapy were selected, with ages ranging from 18 to 85 years old. All enrolled patients had peripheral blood drawn within one week before treatment, and at 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months after treatment for the detection of SHOX2/PTGER4 methylation in plasma circulating tumor DNA (ctDNA).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The median lead time of SHOX2/PTGER4 methylation compared with traditional methods (tumor markers, imaging) for prediction. | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: SHOX2/PTGER4 Methylation Detection Kit (PCR Fluorescence Method).
Disease-free survival: Differences in DFS based on methylation status after treatment. | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: Kaplan-Meier method.
Dynamic concentration changes: The relative change rate of methylation levels before and after treatment and during recurrence. | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: SHOX2/PTGER4 Methylation Detection Kit (PCR Fluorescence Method).

SECONDARY OUTCOMES:
The rate of methylation "turning negative" after treatment | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: SHOX2/PTGER4 Methylation Detection Kit (PCR Fluorescence Method).
The relationship between methylation status and overall survival. | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: Multivariate Cox regression, Log-rank test
Forecast performance | Through study completion, an average of 2 years.
  Measure time point of outcome: Preoperatively, 3 days, 1 month, 3 months, 6 months, 12 months, 18 months and 24 months postoperatively, and at the time of recurrence.
  Measure method: Receiver Operating Characteristic Curve.

CONTACTS AND LOCATIONS:
Overall Officials: Yuqing Huang, Principal Investigator — Beijing Haidian Hospital
Locations (1):
- Beijing Haidian Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No